CLINICAL TRIAL: NCT00441623
Title: A Single Centre Observational Cohort Study on the Prognostic Relevance of P-cresol and Related Uremic Retention Solutes in the Development and/or Progression of Renal Failure and Cardiovascular Disease in Chronic Kidney Disease Patients
Brief Title: The Role of P-cresol and Related Protein Fermentation Metabolites in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Björn Meijers, Prof, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: PCS001
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; cardiovascular disease; risk stratification
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma Urine (if provided by patient)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: observational — effect of protein-bound uremic retention solutes

SUMMARY:
Study on the natural history of uremic retention solutes in patients with mild-to-moderate chronic kidney disease

DETAILED DESCRIPTION:
Protein-bound uremic retention solutes are increasingly recognized to play a role in the pathophysiology of the uremic syndrome. Numerous in vitro findings are indicative for their implication in the biochemical and physiological changes of uremia. Several of these protein-bound retention solutes originate from bacterial protein fermentation in the colon. p-cresyl sulfate, a fermentation metabolite of the amino acid tyrosine, is considered a prototype of this group of uremic solutes. The protein binding of this molecule was shown to be about 90% in end-stage renal disease patients. Several data have suggested that p-cresol plays a role in the immunodeficiency of uremia. Recently, a link between the molecule and endothelial dysfunction has been demonstrated. Also other members of the class of protein-bound solutes have been found to be associated with immune dysfunction, endothelial cell dysfunction and, closely related to the latter, oxidative stress.

Free serum levels of p-cresol were shown to be greater in stage 5 chronic kidney disease (CKD) patients treated with hemodialysis (HD) hospitalized for infectious disease. Furthermore, a positive relationship was found between serum total p-cresol level and a uremic symptom score in patients treated with peritoneal dialysis (PD), whereas a correlation with small water-soluble solutes and the middle molecule β2-microglobulin was absent. A recent prospective observational study in stage 5 CKD patients treated with conventional HD (3 x 4 hours per week) indicated that the accumulation of p-cresol is a risk factor for overall mortality.

Data on the serum concentrations of p-cresol in chronic kidney disease patients are lacking. The investigators hypothesise that the serum concentration of p-cresol is an independent predictor of progression to end stage renal disease and is an independent predictor for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Chronic kidney disease, stage 1-4 kDOQI

Exclusion criteria

* age below 18
* Kidney transplant recipient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chronic kidney disease patients KDOQI stage 1-5 not yet on dialysis
Sampling Method: Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2005-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Björn KI Meijers, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Pieter Evenepoel, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evenepoel P, Claes K, Viaene L, Bammens B, Meijers B, Naesens M, Sprangers B, Kuypers D. Decreased Circulating Sclerostin Levels in Renal Transplant Recipients With Persistent Hyperparathyroidism. Transplantation. 2016 Oct;100(10):2188-93. doi: 10.1097/TP.0000000000001311. PMID 27379556
- [Derived] Evenepoel P, Meijers B, Viaene L, Bammens B, Claes K, Kuypers D, Vanderschueren D, Vanrenterghem Y. Fibroblast growth factor-23 in early chronic kidney disease: additional support in favor of a phosphate-centric paradigm for the pathogenesis of secondary hyperparathyroidism. Clin J Am Soc Nephrol. 2010 Jul;5(7):1268-76. doi: 10.2215/CJN.08241109. Epub 2010 May 6. PMID 20448073
- [Derived] Meijers BK, Claes K, Bammens B, de Loor H, Viaene L, Verbeke K, Kuypers D, Vanrenterghem Y, Evenepoel P. p-Cresol and cardiovascular risk in mild-to-moderate kidney disease. Clin J Am Soc Nephrol. 2010 Jul;5(7):1182-9. doi: 10.2215/CJN.07971109. Epub 2010 Apr 29. PMID 20430946